CLINICAL TRIAL: NCT02592226
Title: Clinical Significance of Alveolar Recruitment Maneuver During Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-PP-11
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2015-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Procedure: Anesthesia: standardized
- Protocol Group (Experimental)
  Interventions: Procedure: Anesthesia: alveolar recruitment maneuver

INTERVENTIONS:
Procedure: Anesthesia: alveolar recruitment maneuver
  Arms: Protocol Group
Procedure: Anesthesia: standardized
  Arms: Control group

SUMMARY:
The ventilation of the patient under general anesthesia is an old problem and extensively studied, especially in visceral surgery, higher risk of postoperative complications. Studies have recently shown the impact of a lung-protective ventilation in visceral surgery, however obese patients are often excluded, and alveolar recruitment maneuver has never been studied independently.

The investigators are conducting a randomized controlled prospective study to investigate the clinical value to achieve alveolar recruitment maneuver routinely in patients undergoing bariatric surgery.

The objective is to show the reduction in dyspnea, oxygen dependency: reflection of atelectasis and the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients surgery for bariatric surgery (sleeve, gastric bypass, gastric banding ablation)
* planned surgery,
* ASA 1-2-3,

Exclusion Criteria:

* Severe COPD
* Severe emphysema,
* Pneumothorax,
* Right sided heart failure,
* Severe heart failure
* Emergency surgery,
* ASA 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
occurrence of dyspnea | 2 hours
oxygen saturation | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde SEVERAC, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Severac M, Chiali W, Severac F, Perus O, Orban JC, Iannelli A, Debs T, Gugenheim J, Raucoules-Aime M. Alveolar recruitment manoeuvre results in improved pulmonary function in obese patients undergoing bariatric surgery: a randomised trial. Anaesth Crit Care Pain Med. 2021 Jun;40(3):100775. doi: 10.1016/j.accpm.2020.09.011. Epub 2020 Nov 1. PMID 33137453